CLINICAL TRIAL: NCT01522092
Title: The Effect of Escitalopram on Exacerbation Rates and Quality of Life in Patients With Anxiety Associated With Severe COPD
Brief Title: Escitalopram in Anxiety Associated Chronic Obstructive Pulmonary Disease (COPD) Exacerbations
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Study was not given ethical approval- a alternative protocol required
Sponsor: Hull University Teaching Hospitals NHS Trust (Other Government)
Responsible Party: Principal Investigator, Prof A H Morice, professor of Respiratory Medicine, Hull University Teaching Hospitals NHS Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Escit160710; 2010-022038-10 (EudraCT Number)
Record Dates: First submitted 2012-01-27; First posted 2012-01-31 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2017-03

CONDITIONS: Anxiety; COPD
Keywords: Exacerbations
MeSH Terms: conditions — Anxiety Disorders; Pulmonary Disease, Chronic Obstructive | interventions — Escitalopram; Dexetimide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- escitalopram (Experimental): escitalipram tablets 5mg, 10 mg and 20 mg, once a day for 12 months
  Interventions: Drug: escitalopram

INTERVENTIONS:
Drug: escitalopram — 5mg-20mg, tablet, od, 12 months
  Other Names: Cipralex

SUMMARY:
Anxiety and depression are common in patients with severe chronic obstructive pulmonary disease (COPD). Frequently exacerbation's of breathlessness are associated with panic/fear and indeed this may be the main cause for the for hospital admission. Patients prone to a tendency to experience and communicate somatic distress in response to psychosocial stress and to seek medical help for it are top of the "frequent flyer" league, costing the health care economy dearly. This is a particular problem in Hull with the high levels of smoking and urban deprivation combining to place the city at the bottom of the Department of Health COPD league tables.

Our hypothesis is that an effective treatment for anxiety will reduce the number of episodes of hospital admission by reducing the panic/fear element of mild COPD exacerbation's thus allowing the patient time to access the existing community based support services.

ELIGIBILITY:
Inclusion Criteria:

* Male/females aged between 40-80 years.
* Previous diagnosis of COPD confirmed by the GOLD criteria.
* At least two previous admissions to hospital for acute exacerbation of COPD.
* Physician diagnosed anxiety
* At least Mild anxiety score on HADS and GAD-7
* On a stable therapeutic regimen for COPD for 8 weeks prior to inclusion
* Known history of cigarette smoking at least 10 pack yrs
* Willing and able to comply with study procedures
* Able to provide written informed consent to participate

Exclusion Criteria:

* Current or past diagnosis of asthma
* Long-term oxygen therapy
* Currently on treatment with anti-depressives
* Serious inter-current illness (eg lung cancer)
* One year survival considered unlikely
* Patients who have evidence of alcohol or drug abuse
* Participation in another clinical trial with an investigational drug in four weeks preceding the screening visit
* Clinically significant or unstable concurrent disease e.g. left ventricular failure, diabetes mellitus
* Known or suspected hypersensitivity to escitalopram

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
exacerbation rate | 12 months
  comparison of the rate of COPD exacerbation in the year preceding treatment with that on escitalopram treatment in patients with COPD adjudged to have a significant element of anxiety.

SECONDARY OUTCOMES:
Quality of life | 12 months
  To assess the effect of escitalopram on the patient's quality of life, as measured by St Georges Respiratory Questionnaire
Hospital Anxiety and depression scale (HADS) | 12 months
  Change in HADS score at 3, 9, and 12 months from baseline
General anxiety disorder(GAD-7) | 12 months
  Change in GAD-7 score at 3,9 and 12 months from baseline
Modified Medical Research Council (MMRC) dyspnoea scale | 12 month
  Change in Modified Medical research council Dyspnoea scale at 3, 9 and 12 months from baseline
BODE index | 12 months
  Change in BODE index at 3, 9 and 12months from baseline
Health related utilisation | 12 months
  Number of health related utilisations from baseline to 3, 9 and 12 months
Spirometry | 12 months
  Change in Forced expired volume in 1 sec, Forced vital capacity and Peak expiratory flow measured at 3, 9 and 12 months from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Alyn H Morice, Professor, Principal Investigator — Hull University Teaching Hospitals NHS Trust
Locations (1):
- Respiratory Medicine, Clinical trials Unit, Castle Hill Hospital, Cottingham, East Yorkshire, United Kingdom